CLINICAL TRIAL: NCT05002127
Title: A Phase 2/3 Study of Evorpacept (ALX148) in Patients With Advanced HER2-Overexpressing Gastric/Gastroesophageal Junction Adenocarcinoma (ASPEN-06)
Brief Title: A Study of Evorpacept (ALX148) in Patients With Advanced HER2+ Gastric Cancer (ASPEN-06)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALX Oncology Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT148006
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Gastric Adenocarcinoma
Keywords: ALX148; CD47; SIRPα; Gastric; Gastroesophageal; GEJ; HER2 positive; Ramucirumab; Evorpacept
MeSH Terms: conditions — Stomach Neoplasms | interventions — ALX148; Trastuzumab; Ramucirumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 2 is Open Label; Phase 3 is blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 2 - Arm A (Experimental): Evorpacept (ALX148) 30 mg/kg every two weeks (Q2W) intravenous (IV), trastuzumab (initial dose of 6 mg/kg followed by 4 mg/kg) Q2W IV, ramucirumab 8 mg/kg Q2W IV, and paclitaxel 80 mg/m2 IV Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Evorpacept (ALX148); Drug: Trastuzumab; Drug: Ramucirumab; Drug: Paclitaxel
- Phase 2 - Arm B (Active Comparator): Trastuzumab (initial dose of 6 mg/kg followed by 4 mg/kg) Q2W IV, ramucirumab 8 mg/kg Q2W IV, and paclitaxel 80 mg/m2 IV Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Trastuzumab; Drug: Ramucirumab; Drug: Paclitaxel
- Phase 3 - Arm A (Experimental): Evorpacept (ALX148) 30 mg/kg Q2W IV, trastuzumab (initial dose of 6 mg/kg followed by 4 mg/kg) Q2W IV, ramucirumab 8 mg/kg Q2W IV, and paclitaxel 80 mg/m2 IV Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Evorpacept (ALX148); Drug: Trastuzumab; Drug: Ramucirumab; Drug: Paclitaxel
- Phase 3 - Arm B (Active Comparator): Ramucirumab 8 mg/kg Q2W IV and paclitaxel 80 mg/m2 IV Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Evorpacept (ALX148) — IV Q2W
  Arms: Phase 2 - Arm A; Phase 3 - Arm A
Drug: Trastuzumab — IV Q2W
  Other Names: Herceptin
  Arms: Phase 2 - Arm A; Phase 2 - Arm B; Phase 3 - Arm A
Drug: Ramucirumab — IV Q2W
  Other Names: Cyramza
Drug: Paclitaxel — IV Days 1, 8, and 15 of a 28-day cycle
  Other Names: Taxol

SUMMARY:
A Phase 2/3 Study of Evorpacept (ALX148) in Combination With Trastuzumab, Ramucirumab, and Paclitaxel in Patients With Advanced HER2-overexpressing gastric/GEJ adenocarcinoma.

DETAILED DESCRIPTION:
This is a randomized phase 2 (open-label) / 3 (blinded), international, multi-center study of patients with metastatic HER2-overexpressing gastric/GEJ adenocarcinoma that has progressed on or after prior HER2-directed therapy and fluoropyrimidine- or platinum-containing chemotherapy and are suitable for chemotherapy (2nd-line or 3rd-line). Approximately 450 adult patients are expected to be enrolled in the study across both phases.

The Sponsor has decided not to proceed with the Phase 3 portion of the study due to strategic considerations.

ELIGIBILITY:
Inclusion Criteria:

* HER2-overexpressing advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma that has progressed on or after a prior HER2-directed agent and fluoropyrimidine- or platinum-containing chemotherapy (2nd-line or 3rd-line)
* Adequate Bone Marrow Function.
* Adequate Renal & Liver Function.
* Adequate Performance Status

Exclusion Criteria:

* Patients with known symptomatic central nervous system (CNS) metastases or leptomeningeal disease requiring steroids.
* Prior treatment with any anti-CD47 or anti-SIRPα agent.
* Prior treatment with ramucirumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase 2 | Last randomized patient on study at least 16 weeks
  Percentage of patients with objective response per RECIST 1.1
Phase 3 | From the date of randomization to the date of death (due to any cause), up to 36 months postdose
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (83):
- United States (5):
  - The Oncology Institute of Hope & Innovation, Anaheim, California
  - University of California Los Angeles, Los Angeles, California
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - NEXT Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Icon Cancer Centre Southport, Southport, Queensland
  - Monash Medical Centre, Clayton, Victoria
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Czechia (3):
  - Fakultní Nemocnice Hradec Králové, Hradec Králové
  - Fakultní Nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice v Praze, Prague
- France (9):
  - Centre Hospitalier Régional et Universitaire de Besançon - Hôpital Jean-Minjoz, Besançon
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Hôpital Morvan, Brest
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hôpital Saint-Antoine, Paris
  - Hôpital Trousseau, Paris
  - Hôpital Rangueil, Toulouse
- Italy (5):
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione Garibaldi, Catania
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Azienda Sanitaria Universitaria Friuli Centrale - P.O. Santa Maria della Misericordia, Udine
- Japan (15):
  - National Cancer Center Hospital East, Chiba
  - Kyushu Cancer Center, Fukuoka
  - Gifu University Hospital, Gifu
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osaka
  - Oita University Hospital - Hasama Campus, Ōita
  - Saitama Cancer Center, Saitama
  - Tohoku University Hospital, Sendai
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Icon Cancer Centre Farrer Park, Singapore
- South Korea (19):
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Hallym University Sacred Heart Hospital, Dongan
  - National Cancer Center - Korea, Goyang-si
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea Saint Vincent's Hospital, Suwon
- Spain (10):
  - Hospital General Universitario de Elche, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Quirónsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (7):
  - Koo Foundation Sun Yat-Sen Cancer Center, Beitou
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital - Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Royal Free Hospital, London
  - Guy's and Saint Thomas' NHS Foundation Trust, London
  - The Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: No